CLINICAL TRIAL: NCT03188211
Title: Simulation-based Technologies to Improve the Appropriate Use of Oral Anticoagulants in Hospitalized Elderly Patients With Atrial Fibrillation
Brief Title: E-learning to Improve Oral Anticoagulant Use in Hospitalized Older People With AF
Acronym: SIM-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BMS ISR # CV185-483
Record Dates: First submitted 2017-06-05; First posted 2017-06-15 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Simulation Training; Anticoagulant Drugs; Elderly; Atrial Fibrillation; Drug Prescriptions; Internal Medicine; Geriatrics
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): Clinicians allocated to intervention arm will receive an e-learning educational program based on simulation-based technologies (Dr Sim). Dr Sim provides a powerful editing system that allows to create clinical cases according to the educational need and purposes. It will be distributed on an e-learning platform, allowing the user to act in a highly interactive learning environment. Management of the virtual patients is carried out interactively and each diagnostic and or therapeutic choice will be supported by any scientific data, guidelines recommendations, drug descriptions and literature references useful to address the best choice for that specific patient as it should be in real practice.
  Interventions: Other: E-learning educational program
- Control (Other): Clinicians allocated to control arm will not receive the e-learning educational program based on simulation-based technologies (Dr Sim).
  Interventions: Other: Control

INTERVENTIONS:
Other: E-learning educational program — A number of 10 cases of patients 65 years of age or older with AF, acutely admitted to Internal Medicine or Geriatric wards for any medical condition, will be edited into the Dr. Sim system. Diagnostic and therapeutic choices for ordinary and/or complex medical situations will be taken through the development of the simulated scenario.
  Other Names: Dr Sim
  Arms: Intervention
Other: Control — Any educational program will be delivered to clinicians assigned to control arm
  Arms: Control

SUMMARY:
Atrial Fibrillation (AF) is the most common cardiac arrhythmia and the main cause of cardioembolic stroke. Oral Anticoagulation (OAC) has been shown to significantly prevent AF-related thromboembolism, however, despite convincing evidences and current guidelines recommendations, OAC tends to be underused in clinical practice especially in the oldest. Education and training to appropriately select people suitable for OAC for stroke prevention could be pivotal in the decision making process. According to the study project, physicians working in Internal Medicine and Geriatric wards, where are mainly admitted elderly people with AF, will undergo to a program of e-learning through computer-based simulation method reproducing clinical scenarios of patients aged 65 years or older, with known or newly diagnosed AF, admitted to hospital for any medical reason and requesting that a decision about long-term antithrombotic therapy is taken.

Primary objective of the study is to investigate whether such educational intervention will improve the appropriate use and prescription rate of OAC in hospitalised elderly patients with AF, multimorbidity and polypharmacy, in comparison to the usual practice.

The study will be a cluster randomised controlled trial involving a network of Internal Medicine and Geriatrics wards. Thirty-two wards will be recruited based on voluntary participation and randomised to receive an educational intervention through computer-based simulation, (N=16) or to continue with the usual practice (N=16). Subjects receiving the intervention will be all the staff physicians of the wards randomised in the intervention arm.

The impact of the intervention compared with the usual practice will be evaluated in patients aged 65 years or older admitted to the participating centres with a known diagnosis of AF or newly diagnosed with AF during the hospitalisation.

ELIGIBILITY:
Inclusion Criteria:

* subjects 65 years of age or older, with known or newly diagnosed AF, admitted to the Internal Medicine and Geriatric wards of the REPOSI network,
* consent to participate to the study.

Exclusion Criteria:

* consent denial to participate to the study,
* absolute contraindication to OAC,
* re-hospitalisation for the subject already included in the study,
* life expectancy less than 6 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 247 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Elderly with AF prescribed with OAC | through study completion, up to 1 year
  difference in the proportion of elderly patients with AF prescribed with OAC between the post-intervention and the pre-intervention observational phase

SECONDARY OUTCOMES:
Number of access to Dr Sim | 1 month
  average number of access to Dr. Sim among the phsyicians of the centres randomised to the intervention during the 1 month intervention phase
Total duration of connection to Dr Sim | 1 month
  average total duration of connection to Dr. Sim among the phsyicians of the centres randomised to the intervention during the 1 month intervention phase
Elderly patients with AF prescribed with any antiplatelet agent | through study completion, up to 1 year
  difference in the proportion of elderly patients with AF prescribed with any antiplatelet agent (and not OAC) between the post-intervention and the pre-intervention observational phase
Elderly patients with AF newly prescribed with OAC agents | through study completion, up to 1 year
  difference in the proportion of elderly patients with AF prescribed with new OAC agents between the post-intervention and the pre-intervention observational phase
Patients experiencing any cerebro or cardiovascular events | 6 month follow up
  proportion of patients experiencing any stroke, transient ischaemic attack (TIA), other major arterial or venous thromboembolism during the 6 months after the hospital discharge
Re-hospitalization rate | 6 month follow up
  proportion of patients re-hospitalised for any cause during the 6 months after the hospital discharge
Minor bleeding events | 6 month follow up
  proportion of patients experiencing a minor bleeding event during the 6 months after hospital discharge)
Major bleeding event | 6 month follow up
  proportion of patients experiencing a major bleeding event during the 6 months after hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Santalucia, MD, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano
Locations (20):
- Italy (20):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna, Bo
  - Istituto Fondazione Poliambulanza, Brescia, BS
  - Policlinico Universitario Mater Domini, Catanzaro, CZ
  - AO Universitaria Policlinico di Modena, Modena, Italia
  - Azienda Ospedaliera S. Gerardo di Monza, Monza, MB
  - Ospedale degli Infermi, Rivoli, TO
  - Azienda Ospedaliera Universitaria - Ospedale Riuniti, Trieste, TS
  - A.O. Ospedale di Circolo e Fondazione Macchi, Varese, VA
  - Azienda Consorziale Ospedaliera Policlinico, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria "Policlinico Vittorio Emanuele", Catania
  - Azienda Ospedaliera Universitaria San Martino - IST, Genoa
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico P. Giaccone, Palermo
  - Azienda SocioSanitaria Territoriale, Ospedale Civile "C.Mira" di Casorate Primo, Pavia
  - Policlinico San Matteo, Pavia
  - Ospedale San Giovanni Calibita Fatebenefratelli, Roma
  - Policlinco Universitario Agostino Gemelli, Rome
  - Ospedale SS Annunziata, Sassari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Proietti M, Antoniazzi S, Monzani V, Santalucia P, Franchi C; SIM-AF Investigators; Fenoglio LM, Melchio R, Fabris F, Sartori MT, Manfredini R, De Giorgi A, Fabbian F, Biolo G, Zanetti M, Altamura N, Sabba C, Suppressa P, Bandiera F, Usai C, Murialdo G, Fezza F, Marra A, Castelli F, Cattaneo F, Beccati V, di Minno G, Tufano A, Contaldi P, Lupattelli G, Bianconi V, Cappellini D, Hu C, Minonzio F, Fargion S, Burdick L, Francione P, Peyvandi F, Rossio R, Colombo G, Monzani V, Ceriani G, Lucchi T, Brignolo B, Manfellotto D, Caridi I, Corazza GR, Miceli E, Padula D, Fraternale G, Guasti L, Squizzato A, Maresca A, Liberato NL, Tognin T, Rozzini R, Bellucci FB, Muscaritoli M, Molfino A, Petrillo E, Dore M, Mete F, Gino M, Franceschi F, Gabrielli M, Perticone F, Perticone M, Bertolotti M, Mussi C, Borghi C, Strocchi E, Durazzo M, Fornengo P, Dallegri F, Ottonello LC, Salam K, Caserza L, Barbagallo M, Di Bella G, Annoni G, Bruni AA, Odetti P, Nencioni A, Monacelli F, Napolitano A, Brucato A, Valenti A, Castellino P, Zanoli L, Mazzeo M. Use of oral anticoagulant drugs in older patients with atrial fibrillation in internal medicine wards. Eur J Intern Med. 2018 Jun;52:e12-e14. doi: 10.1016/j.ejim.2018.04.006. Epub 2018 Apr 12. No abstract available. PMID 29657108
- [Derived] Antoniazzi S, Ardoino I, Proietti M, Monzani V, Mannucci PM, Nobili A, Franchi C; SIM-AF Collaborators. Appropriateness of prescription of oral anticoagulant therapy in acutely hospitalized older people with atrial fibrillation. Secondary analysis of the SIM-AF cluster randomized clinical trial. Br J Clin Pharmacol. 2019 Sep;85(9):2134-2142. doi: 10.1111/bcp.14029. Epub 2019 Jul 19. PMID 31218738
- [Derived] Franchi C, Antoniazzi S, Ardoino I, Proietti M, Marcucci M, Santalucia P, Monzani V, Mannucci PM, Nobili A; SIM-AF Collaborators. Simulation-Based Education for Physicians to Increase Oral Anticoagulants in Hospitalized Elderly Patients with Atrial Fibrillation. Am J Med. 2019 Aug;132(8):e634-e647. doi: 10.1016/j.amjmed.2019.03.052. Epub 2019 May 8. PMID 31075225
- See also: Letters to Editor — http://www.ncbi.nlm.nih.gov/pubmed/29657108